CLINICAL TRIAL: NCT02959918
Title: An Open Label Phase II Multiple Dose Safety, Pharmacokinetic and Pharmacodynamics Study of SEL-212 Followed by Open Label Administration of SEL-037 in Subjects With Symptomatic Gout and Elevated Blood Uric Acid
Brief Title: Multi-Dose Safety/Pharmacodynamic Study of SEL-212/SEL-037 in Subjects With Symptomatic Gout & Elevated Blood Uric Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL-212/201
Record Dates: First submitted 2016-11-06; First posted 2016-11-09 (Estimated); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Gout Chronic; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (14):
- SEL-037 Pegadricase LD (low dose) alone (Experimental): Pegadricase 0.2 mg/kg intravenous (IV) every 28 days for 5 treatments
  Interventions: Drug: SEL-037
- SEL-037 Pegadricase HD (high dose) alone (Experimental): Pegadricase 0.4 mg/kg intravenous (IV) every 28 days for 5 treatments
  Interventions: Drug: SEL-037
- SEL-212, Pegadricase LD & SEL-110 (1a) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.05 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.2 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (1b) (Experimental): Pegadricase 0.4 mg/kg IV plus SEL-110 0.05 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.4 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase LD & SEL-110 (2a) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.08 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.2 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (2b) (Experimental): Pegadricase 0.4 mg/kg IV plus SEL-110 0.08 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.4 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (3a) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.1 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.2 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (3b) (Experimental): Pegadricase 0.4 mg/kg IV plus SEL-110 0.1 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.4 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (4a) (Experimental): Pegadricase 0.4 mg/kg IV plus SEL-110 0.125 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.4 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (4b) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.15 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.2 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (5a) (Experimental): Pegadricase 0.4 mg/kg IV plus SEL-110 0.15 mg/kg IV every 28 days for 3 treatments, followed by pegadricase 0.4 mg/kg IV every 28 days for 2 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (5b) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.15 mg/kg IV every 28 days for 5 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (6a) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.10 mg/kg IV every 28 days for 1 treatment followed by pegadricase 0.2 mg/kg IV plus SEL-110 0.15 mg/kg IV every 28 days for 4 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)
- SEL-212, Pegadricase HD & SEL-110 (6b) (Experimental): Pegadricase 0.2 mg/kg IV plus SEL-110 0.1 mg/kg IV every 28 days for 5 treatments
  Interventions: Drug: SEL-212; Drug: SVP-rapamycin (SEL-110)

INTERVENTIONS:
Drug: SEL-212 — SEL-212, biologic
  Other Names: Pegadricase plus SVP-rapamycin
  Arms: SEL-212, Pegadricase HD & SEL-110 (1b); SEL-212, Pegadricase HD & SEL-110 (2b); SEL-212, Pegadricase HD & SEL-110 (3a); SEL-212, Pegadricase HD & SEL-110 (3b); SEL-212, Pegadricase HD & SEL-110 (4a); SEL-212, Pegadricase HD & SEL-110 (4b); SEL-212, Pegadricase HD & SEL-110 (5a); SEL-212, Pegadricase HD & SEL-110 (5b); SEL-212, Pegadricase HD & SEL-110 (6a); SEL-212, Pegadricase HD & SEL-110 (6b); SEL-212, Pegadricase LD & SEL-110 (1a); SEL-212, Pegadricase LD & SEL-110 (2a)
Drug: SEL-037 — SEL-037, biologic
  Other Names: Pegadricase
  Arms: SEL-037 Pegadricase HD (high dose) alone; SEL-037 Pegadricase LD (low dose) alone
Drug: SVP-rapamycin (SEL-110) — SVP-rapamycin, biologic
  Other Names: SEL-110
  Arms: SEL-212, Pegadricase HD & SEL-110 (1b); SEL-212, Pegadricase HD & SEL-110 (2b); SEL-212, Pegadricase HD & SEL-110 (3a); SEL-212, Pegadricase HD & SEL-110 (3b); SEL-212, Pegadricase HD & SEL-110 (4a); SEL-212, Pegadricase HD & SEL-110 (4b); SEL-212, Pegadricase HD & SEL-110 (5a); SEL-212, Pegadricase HD & SEL-110 (5b); SEL-212, Pegadricase HD & SEL-110 (6a); SEL-212, Pegadricase HD & SEL-110 (6b); SEL-212, Pegadricase LD & SEL-110 (1a); SEL-212, Pegadricase LD & SEL-110 (2a)

SUMMARY:
This is an open label multicenter study to evaluate the safety and tolerability of multiple doses (3 monthly IV infusions) of SEL-212 ( a combination of pegsiticase (SEL-037) and SVP-rapamycin (SEL-110)) followed by multiple doses (2 monthly IV infusions) of pegsiticase (SEL-037) alone for a total of 5 treatment cycles in subjects with symptomatic gout and hyperuricemia. Additional participants will be treated with multiple doses ( 5 monthly IV infusions) of pegsiticase (SEL-037) alone.

Participants will be monitored for safety endpoints through the 5th treatment cycle plus 30 days .Pharmacokinetic samples will be drawn at pre-determined time points in addition to weekly serum uric acid levels.

DETAILED DESCRIPTION:
This is an open label multicenter study to evaluate the safety and tolerability of multiple doses (3 monthly IV infusions) of SEL-212 ( a combination of pegsiticase ( SEL-037, also known as pegadricase) and SVP-rapamycin (SEL-110)) followed by multiple doses (2 monthly IV infusions) of pegsiticase (SEL-037) alone for a total of 5 treatment cycles in participants with symptomatic gout and hyperuricemia. Additional participants will be treated with multiple doses (5 monthly IV infusions) of pegsiticase (SEL-037) alone.

Uricase is an enzyme that converts uric acid to the readily soluble allantoin that is then excreted and SEL-110 is designed to prevent unwanted anti-drug-antibodies (ADAs) from forming. All participants will be monitored for safety and tolerability to drug throughout the study on a weekly schedule. Pharmacokinetic and pharmacodynamic parameters will at specific timepoints to monitor for continued efficacy. Pharmacodynamic parameters measured include uric acid levels and levels of ADAs.

The study duration per enrolled participant will be approximately 6 months including a 1 month screening period followed by 5 treatment cycles and an end of treatment visit which will occur 30 days after the last IV infusion .

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 21-75 inclusive) men and women of non child bearing potential with established or symptomatic gout which is defined as having at least ONE of any of the 3 following factors:

   1. ≥ 1 tophus
   2. 1 gout flare within the last 6 months
   3. Chronic gouty arthropathy
2. Screening serum uric acid of >6 mg/dL
3. On a gout flare prophylactic regimen for 7 days prior to first dose
4. Willing to provide written informed consent prior to first study procedure is performed.
5. Understands and is willing and able to comply with study requirements, including the schedule of follow-up visits.

Exclusion Criteria:

1. History of anaphylaxis or severe allergic reaction.
2. History of an allergy to pegylated products.
3. Women of child bearing potential, Defined as:

   * <6 weeks after surgical bilateral salpingooperhectony with or without hysterectomy
   * Pre or perimenopausal ( < less than 24 months of natural amenorrhea)
4. Initiation or change in dose of hormone-replacement therapy for menopausal women less than 1 month prior to the Screening Visit or during the Screening Phase would be exclusionary. If after being on a stable dose of hormone-replacement therapy for one month the patient may be considered for the study if she continues to meet all other inclusion and exclusion criteria
5. Uncontrolled diabetes with baseline HbA1c ≥8%;
6. Glucose-6-phosphate dehydrogenase deficiency;
7. Uncontrolled hypertension
8. Ongoing treatment for arrhythmia, including placement of an implantable defibrillator;
9. History of coronary artery disease, including myocardial infarction;
10. Congestive heart failure, New York Heart Association Class III or IV;
11. ECG with evidence of prior myocardial infarction, clinically significant arrhythmia, or other abnormalities that, in the opinion of the investigator, are consistent with significant underlying cardiac disease;
12. History of hematological or autoimmune disorders, is immunosuppressed or immunocompromised;
13. Prior exposure to any experimental or marketed uricase (e.g., rasburicase (Elitek, Fasturtec), pegloticase (Krystexxa®), pegsiticase (SEL-037)
14. History of malignancy within the last 5 years other than basal skin cancer;
15. Subjects who, in the opinion of the investigator, present with a condition that would compromise their safety or that would make study completion unlikely.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Anaheim Clinical Trials, Anaheim, California
  - Tri West Research Associates LLC, El Cajon, California
  - Irvine Center for Clinical Research Inc., Irvine, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Omega Research Consultants LLC, DeBary, Florida
  - Compass Research LLC, Orlando, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Advanced Clinical Research, Boise, Idaho
  - L-MARC, Louisville, Kentucky
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kivitz A, DeHaan W, Azeem R, Park J, Rhodes S, Inshaw J, Leung SS, Nicolaou S, Johnston L, Kishimoto TK, Traber PG, Sands E, Choi H. Phase 2 Dose-Finding Study in Patients with Gout Using SEL-212, a Novel PEGylated Uricase (SEL-037) Combined with Tolerogenic Nanoparticles (SEL-110). Rheumatol Ther. 2023 Aug;10(4):825-847. doi: 10.1007/s40744-023-00546-0. Epub 2023 Apr 17. PMID 37069364

RESULTS

PARTICIPANT FLOW:
Groups:
- SEL-037 (Pegadricase) Low Dose: Pegadricase 0.2 mg/kg IV every 28 days for up to 5 doses
- SEL-037 (Pegadricase) High Dose: Pegadricase 0.4mg/kg IV every 28 days for up to 5 doses
- SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.05 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.05 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.08 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.08 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.125 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 5 doses
- SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low 1 Dose Then SEL-110 0.1 mg/kg + SEL-037 Low for 4 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 1 dose then SEL-110 (0.1 mg/kg) + Pegadricase 0.2 mg/kg every 28 days for 4 doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 5 doses
Period: Overall Study
Arm/Group | SEL-037 (Pegadricase) Low Dose | SEL-037 (Pegadricase) High Dose | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low 1 Dose Then SEL-110 0.1 mg/kg + SEL-037 Low for 4 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses
Started | 3 | 3 | 9 | 10 | 6 | 11 | 11 | 12 | 14 | 13 | 14 | 23 | 11 | 12
Completed | 0 | 0 | 1 | 1 | 1 | 5 | 6 | 6 | 7 | 7 | 8 | 11 | 4 | 6
Not Completed | 3 | 3 | 8 | 9 | 5 | 6 | 5 | 6 | 7 | 6 | 6 | 12 | 7 | 6
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0
Not completed — Stopping Rule Met | 1 | 0 | 3 | 4 | 5 | 3 | 2 | 4 | 1 | 1 | 3 | 5 | 2 | 1
Not completed — Sponsor Decision, Pause in Clinical Trial | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Hospitalized, out of window for next dosing period | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI Discretion due to abnormal Hgb results | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject under-dosed with study drug and removed by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SEL-037 (Pegadricase) Low Dose: Pegardricase 0.2 mg/kg every 28 days for up to 5 doses
- SEL-037 (Pegadricase) High Dose: Pegardricase 0.4 mg/kg every 28 days for up to 5 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low for 1 Dose Then SEL-110 0.1 mg/kg + SEL-037 Low 4 Doses: SEL-212: Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 1 Dose Then SEL-110 0.1 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 4 Doses
- Total: Total of all reporting groups
Arm/Group | SEL-037 (Pegadricase) Low Dose | SEL-037 (Pegadricase) High Dose | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low for 1 Dose Then SEL-110 0.1 mg/kg + SEL-037 Low 4 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses | Total
Number analyzed (Participants) | 3 | 3 | 9 | 10 | 6 | 11 | 11 | 12 | 14 | 13 | 14 | 23 | 11 | 12 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 7 | 9 | 4 | 6 | 10 | 10 | 8 | 12 | 12 | 21 | 11 | 10 | 126
  >=65 years | 0 | 0 | 2 | 1 | 2 | 5 | 1 | 2 | 6 | 1 | 2 | 2 | 0 | 2 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 2 | 1 | 3 | 1 | 0 | 0 | 14
  Male | 3 | 3 | 9 | 9 | 6 | 8 | 10 | 10 | 12 | 12 | 11 | 22 | 11 | 12 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Number Analyzed: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number Analyzed: Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4
  Number Analyzed: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Number Analyzed: Black or African American | 1 | 2 | 2 | 2 | 2 | 2 | 3 | 4 | 2 | 6 | 4 | 7 | 1 | 2 | 40
  Number Analyzed: White | 2 | 0 | 7 | 5 | 4 | 9 | 8 | 8 | 10 | 6 | 10 | 14 | 10 | 10 | 103
  Number Analyzed: Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Multiple Intravenous Infusions of SEL-037 or SEL-212 as Assessed by the Percentage of Participants Experiencing Serious Adverse Events and Those Adverse Events Reported by 5 Percentage or More in the Safety Analysis Set
Description: To determine the safety and tolerability of SEL-037 (pegadricase) after up to 5 monthly infusions, of SEL-212 for 3 monthly infusions followed by 2 monthly infusions of SEL-037 (pegadricase), or of SEL-212 for 5 monthly infusions as assessed by the percentage of participants in a treatment arm experiencing serious adverse events and percentage of participants experiencing those adverse events that were reported by 5 or more percentage of participants in any arm in the safety analysis set
Time Frame: Five monthly infusions
Population: Safety analysis set, dosed subjects
Measure: Count of Participants; unit: Participants
Groups:
- SEL-212: SEL-110(0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037(0.4 mg/kg) for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.05 mg/kg + Pegadricase 0.4 mg/kg every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.08 mg/kg + SEL-037 (pegadricase) 0.2 mg/kg every 28 days for 3 doses followed by SEL-037 0.2 mg/kg every 28 days for 2 doses
- SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low Dose x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low x 4 Doses: SEL-212: Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg x 1 Then SEL-110 0.1 mg/kg + Pegadricase 0.2 mg/kg x 4 Doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses: SEL-212: Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.2 mg/kg every 28 days for 5 doses
Arm/Group | SEL-037 (Pegadricase) Low Dose | SEL-037 (Pegadricase) High Dose | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110(0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037(0.4 mg/kg) for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low Dose x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low x 4 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses
Number analyzed (Participants) | 3 | 3 | 9 | 10 | 6 | 11 | 11 | 12 | 14 | 13 | 14 | 23 | 11 | 12
Participants | 3 | 3 | 9 | 10 | 6 | 11 | 11 | 12 | 14 | 13 | 14 | 23 | 11 | 12

2. Secondary Outcome: Number of Participants With Reduced Serum Uric Acid After Multiple Monthly IV Infusions With or Without SEL-110
Description: Measurement of the number of participants with reduced serum uric acid after multiple monthly infusions with or without SEL-110 as determined by values of sUA < 6 mg/dL at the end of Treatment Period 3 and at the end of Treatment Period 5 in eligible subjects
Time Frame: 3 and 5 months
Population: Eligible subjects are those who received the entire first dose, did not discontinue due to withdrawal of consent (during TP 1-4), a protocol deviation (during TP1-2) or a non-study drug-related SAE (during TP1-2). The outcome data is presented with arms combined by regimen (i.e. SEL-037 alone; SEL-212 for 3 doses & SEL-037 for 2 doses; or SEL-212 for 5 doses) rather than by dosing arm as the outcome is most effected by the SEL-212 combination which results in suppression of anti-drug antibodies.
Measure: Count of Participants; unit: Participants
Groups:
- SEL-037 (Pegadricase): SEL-037 every 28 days for up to 5 doses
- SEL-212 for 3 Doses Followed by SEL-037 for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) + SEL-037 (pegadricase) every 28 days for 3 doses followed by SEL-037 every 28 days for 2 doses
- SEL-212 for 5 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) + SEL-037 (pegadricase) every 28 days for 5 doses
Arm/Group | SEL-037 (Pegadricase) | SEL-212 for 3 Doses Followed by SEL-037 for 2 Doses | SEL-212 for 5 Doses
Number analyzed (Participants) | 3 | 73 | 32
Participants
  Treatment Period 3 | 0 | 51 | 23
  Treatment Period 5 | NA — No subjects in the arm were dosed during treatment period 5 | 27 | 21

3. Secondary Outcome: Number of Participants With Reduced Serum Uric Acid After Multiple Monthly IV Infusions With or Without SEL-110
Description: as for outcome 2
Time Frame: 3 and 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | SEL-037 (Pegadricase) Low Dose | SEL-037 (Pegadricase) High Dose | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110(0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037(0.4 mg/kg) for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low Dose x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low x 4 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses
Number analyzed (Participants) | 2 | 1 | 6 | 5 | 6 | 8 | 10 | 10 | 8 | 9 | 11 | 18 | 6 | 8
Participants
  Treatment Period 3 | 0 | 0 | 2 | 1 | 4 | 6 | 7 | 7 | 7 | 8 | 9 | 12 | 5 | 6
  Treatment Period 5 | NA — No subjects in the arm were dosed during treatment period 5 | NA — No subjects in the arm were dosed during treatment period 5 | 1 | 1 | 0 | 3 | 3 | 4 | 5 | 4 | 6 | 11 | 4 | 6

ADVERSE EVENTS:
Time Frame: 5 months
Groups:
- SEL-037 (Pegadricase) High Dose: Pegadricase 0.4 mg/kg IV every 28 days for up to 5 doses
- SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.05 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.05 mg/kg + Pegadricase 0.4 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.08 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.08 mg/kg + Pegadricase 0.4 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.4 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.125 mg/kg + Pegadricase 0.4 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.2 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.4 mg/kg IV every 28 days for 3 doses followed by Pegadricase 0.4 mg/kg IV every 28 days for 2 doses
- SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 5 doses
- SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low Dose x 4 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.15 mg/kg + Pegadricase 0.2 mg/kg x 1 dose then SEL-110 0.1 mg/kg + Pegadricase 0.2 mg/kg x 4 doses IV every 28 days
- SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses: SEL-212 - Combination of SEL-110 (nanoparticle encapsulating rapamycin) 0.1 mg/kg + Pegadricase 0.2 mg/kg IV every 28 days for 5 doses
Arm/Group | SEL-037 (Pegadricase) Low Dose | SEL-037 (Pegadricase) High Dose | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low Dose x 4 Doses | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 0/10 | 0/6 | 0/11 | 0/11 | 0/12 | 0/14 | 0/13 | 0/14 | 0/23 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/9 | 0/10 | 0/6 | 1/11 | 2/11 | 4/12 | 2/14 | 0/13 | 1/14 | 3/23 | 1/11 | 2/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/9 | 8/10 | 6/6 | 10/11 | 10/11 | 12/12 | 14/14 | 12/13 | 14/14 | 21/23 | 9/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEL-037 (Pegadricase) Low Dose (N=3) | SEL-037 (Pegadricase) High Dose (N=3) | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=9) | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=10) | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=6) | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=12) | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=14) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=13) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=14) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses (N=23) | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low Dose x 4 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses (N=12)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gout flare (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEL-037 (Pegadricase) Low Dose (N=3) | SEL-037 (Pegadricase) High Dose (N=3) | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=9) | SEL-212: SEL-110 (0.05 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=10) | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=6) | SEL-212: SEL-110 (0.08 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=12) | SEL-212: SEL-110 (0.125 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=14) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 3 Doses Then SEL-037 Low Dose for 2 Doses (N=13) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 High Dose for 3 Doses Then SEL-037 High Dose for 2 Doses (N=14) | SEL-212: SEL-110 (0.15 mg/kg) + SEL-037 Low Dose for 5 Doses (N=23) | SEL-212: SEL-110 0.15 mg/kg + SEL-037 Low x 1 Then SEL-110 0.1 mg/kg + SEL-037 Low Dose x 4 Doses (N=11) | SEL-212: SEL-110 (0.1 mg/kg) + SEL-037 Low Dose for 5 Doses (N=12)
Gout flare (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (4) | 2 (3) | 4 (8) | 4 (10) | 6 (15) | 4 (10) | 4 (10) | 8 (23) | 5 (9) | 5 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 4 (4) | 3 (5) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 1 (1) | 4 (5) | 0 (0) | 1 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 3 (5) | 3 (6) | 3 (5) | 1 (2) | 3 (4) | 4 (8) | 3 (8) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (2) | 4 (4) | 3 (4) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (3) | 2 (5) | 1 (2) | 2 (3)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (6) | 3 (4) | 1 (2) | 1 (1) | 2 (3) | 1 (2)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (3) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Oesophageal oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Formication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ejaculation failure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Semen volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic atrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flash (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02959918/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02959918/SAP_001.pdf